CLINICAL TRIAL: NCT03873857
Title: Prospective Multi-Center Observational Study to Assess Effectiveness of Venclexta (Venetoclax) in Population of Relapse or Refractory Chronic Lymphocytic Leukemia Patients in Routine Clinical Practice in Russian Federation (FORTE)
Brief Title: A Study to Assess Effectiveness of Venclexta (Venetoclax) in Patients With Relapse or Refractory Chronic Lymphocytic Leukemia in Routine Clinical Practice in Russian Federation
Acronym: FORTE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-569
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Cancer
Keywords: Chronic Lymphocytic Leukemia (CLL); Cancer; Observational Study; Venetoclax; Relapsed Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — venetoclax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax: Participants in this observational study will receive treatment with venetoclax for up to 24 months for treatment of relapsed or refractory CLL.
  The prescription of a treatment regimen is at the discretion of the physician in accordance with local clinical practice and label, is made independently from this observational study and precedes the decision to offer the patient the opportunity to participate in this study.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — tablet;oral
  Other Names: Venclexta; ABT-199

SUMMARY:
This study seeks to assess the effectiveness and safety of venetoclax in patients with relapsed and refractory chronic lymphocytic leukemia (CLL) in a real-world setting across clinical practice in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of relapsed or refractory CLL.
* Patient for whom the physician has decided to initiate CLL treatment with venetoclax (mono and combo therapy), or up to 4 weeks after venetoclax treatment initiation
* Patient voluntarily agrees to participate in this study and signs informed consent form

Exclusion Criteria:

* Has contraindications to venetoclax as listed on the approved local label in Russian Federation.
* Has Richter syndrome
* Participated in a clinical trial with an investigative drug for CLL within 30 days prior to treatment initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed or refractory CLL in a real-world clinical practice setting.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) 12 Months after Treatment Initiation | Up to approximately 12 months after treatment initiation
  ORR is defined as the percentage of participants who reach either complete remission (CR), CR with incomplete bone marrow recovery (CRi), nodular partial remission (nPR), or partial remission (PR) to treatment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) 24 Months after Treatment Initiation | Up to approximately 24 months after treatment initiation
  ORR is defined as the percentage of participants who reach either complete remission (CR), CR with incomplete bone marrow recovery (CRi), nodular partial remission (nPR), or partial remission (PR) to treatment.
Time to First Response to Treatment | Up to approximately 24 months
  The time to response to treatment is defined by the time between the date of the first venetoclax intake and the date of the first assessment having documented a response (CR, CRi, nPR, and PR).
Time to Best Response to Treatment | Up to approximately 24 months
  The time to best response to treatment is defined by the time between the date of the first venetoclax intake and the date of the best response documented (CR, CRi, nPR, and PR).
Duration of Response (DoR) | Up to approximately 24 months
  DoR defined as the number of days from the date of first response (CR, CRi, nPR, or PR) to the date of disease progression or death from any cause, whichever comes first.
Time To Next Treatment | Up to approximately 24 months
  The time to next treatment is defined as the time between the date of the first venetoclax intake and the date of the first next treatment intake after venetoclax discontinuation.
Percentage of Patients with Undetectable Minimal Residual Disease (MRD) | Up to approximately 24 months
  Patients will be defined as having a clinical remission in the absence of MRD when they have blood or marrow with less than one CLL cell per 10000 leucocytes.
Overall Survival (OS) Rate | Up to approximately 24 months
  OS is defined as number of days from the date of first dose to the date of the observational period end or death for all dosed patients.
Progression-free Survival (PFS) | Up to approximately 24 months
  Progression-free survival is defined as the interval between the first treatment day to the first sign of disease progression or death from any cause
Change from Baseline in RAND Short Form (SF)-36 Questionnaire | Up to approximately 24 months
  Patient quality of life was measured by the RAND-36 health-related quality of life (HRQoL) survey instrument. This questionnaire is comprised of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (20):
- Russia (20):
  - Oncology Dispensary #2 /ID# 215831, Sochi, Krasnodarskiy Kray
  - Moscow State budget healthcare /ID# 212875, Moscow, Moscow
  - Moscow Regional Research and Clinical Institute n.a. Vladimirskiy (MONIKI) /ID# 215830, Moscow, Moscow Oblast
  - Academician I.P. Pavlov First St. Petersburg State Medical University /ID# 212368, Saint Petersburg, Sankt-Peterburg
  - Central City Hospital #7 /ID# 212373, Yekaterinburg, Sverdlovsk Oblast
  - Regional Children's Clinical Hospital of Volgograd /ID# 212366, Volgograd, Volgograd Oblast
  - Krai Clinical Hospital /ID# 224952, Barnaul
  - GBUZ Regional Cancer center /ID# 216871, Irkutsk
  - Krai Clinical Hospital #1 /ID# 212367, Khabarovsk
  - Kirov Regional Clinical Hospital /ID# 217579, Kirov
  - Policlinic #2 /ID# 214778, Oryol
  - Clinical Medico-Sanitary Unit #1 /ID# 212364, Perm
  - Russian Research Institute of Hematology and Transfusiology of the FMBA /ID# 212372, Saint Petersburg
  - Almazov National Medical Research Centre /ID# 212365, Saint Petersburg
  - Komi Republican Oncology Dispensary /ID# 212370, Syktyvkar
  - City Clinical Hospital # 5 /ID# 212369, Vladimir
  - Regional Clinical Hospital of Vologda /ID# 212471, Vologda
  - Republican Hospital #1 - National Center of Medicine of Sakha (Yakutia) /ID# 212371, Yakutsk
  - Sverdlovsk Regional Clinical Hospital #1 /ID# 214777, Yekaterinburg
  - Sakhalin Regional Clinical Hospital /ID# 222503, Yuzhno-Sakhalinsk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P19-569#additional-resources-section